CLINICAL TRIAL: NCT00246194
Title: The SOURCE Study: Schizophrenia Outcomes-utilization, Relapse, and Clinical Evaluation: a Prospective 2-year Observational Study of Patients With Schizophrenia Who Initiate Treatment With Injectable Risperidone Long-acting Microspheres (RISPERDAL CONSTA)
Brief Title: Observational Study in Patients With Schizophrenia Treated With Long-Acting Risperidone Injection (RISPERDAL CONSTA)
Acronym: SOURCE
Status: Completed | Type: Observational
Sponsor: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: CR005035; RIS-OUT-173 (Other: Janssen, LP); RISSCH4001 (Other: Janssen, LP); NCT01571154 (obsolete NCT alias)
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mental disorder; DSM-IV; RISPERDAL CONSTA; Risperidone; Long-acting risperidone; Disorganized; Catatonic; Paranoid
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Catatonia | interventions — Risperidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with schizophrenia: Long-acting injectable of risperidone given as per the prescription from the prescribing physician (Observational study).
  Interventions: Drug: risperidone (RISPERDAL CONSTA)

INTERVENTIONS:
Drug: risperidone (RISPERDAL CONSTA) — Long-acting injectable of risperidone given as per the prescription from the prescribing physician.
  Other Names: RISPERDAL CONSTA

SUMMARY:
The purpose of this study is to examine treatment practices of adult schizophrenia patients by their own doctors, and to assess patient outcomes when treated with long-acting risperidone injection over a two-year period of observation.

DETAILED DESCRIPTION:
This is a 2-year, prospective (a study in which the patients are identified and then followed forward in time for the outcome of the study), multi-center (at multiple sites), longitudinal (study that involves repeated observations of the same outcomes in the same people over long periods of time), observational study (study in which the investigators/ physicians observe the patients and measure their outcomes) in adults with schizophrenia (mental disorder characterized by a breakdown of thought processes and by poor emotional responsiveness). Physicians will determine the appropriate treatment for their patients, according to their usual practice. Patients starting treatment with long-acting risperidone injection (an antipsychotic medication) and meeting all the study criteria will be enrolled in the study. They will receive a dose of 25, 37.5 or 50 mg of risperidone every 2 weeks by intramuscular injection, and continue their treatment for schizophrenia according to usual care by their physicians. Patients will be asked questions at baseline and every three months for a period of two years to assess: efficacy of the medication, how well the patient is functioning, use of healthcare resources (eg, emergency room visits and hospitalizations) patient work status, quality of life and patient satisfaction with the medicine. Safety will be monitored throughout the study duration of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients had schizophrenia (disorganized, catatonic, paranoid, residual, or undifferentiated) that met disease diagnostic criteria as defined in Diagnostic and Statistical Manual of Mental Disorders IV ([DSM-IV]
* Requiring new treatment with long-acting risperidone injectable
* Patients were cooperative, reliable, and able to complete all aspects of the protocol

Exclusion Criteria:

* Use of an investigational drug in the past 30 days
* At risk to self or others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2004-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 24 months in Clinical Global Impression of Severity (CGI-S) scores | Baseline (Month 0) to 24 months
  The CGI-S is a 7-point scale ranging from 1 to 7 (normal, not at all ill to among the most severely ill patients), which measures disease severity in psychiatric patients. The scale is completed by physician.
Clinical Global Impression of Change (CGI-C) scores during 24 months | 24 months
  The CGI-C is a 7-point scale ranging from 1 to 7 (very much improved to very much worse), which is used to rate the change in the patient's illness compared to baseline. The scale assesses the patient's improvement over time. The scale is completed by physician.
Change from baseline to 24 months in Global Assessment of Function (GAF) scores | Baseline to 24 months
  GAF is completed by the physician. GAF is a single item rating of the patient's psychological, social, and occupational functioning on a hypothetical continuum of mental health-illness. Respondents are asked to rate the subject's lowest level of functioning in the last week. GAF scores range from 0 to 100. (0 = Inadequate information, 1 = Persistent danger of severely hurting self or others and 100 = Superior functioning in a wide range of activities).
Change from baseline to 24 months in Personal and Social Performance (PSP) scores | Baseline to 24 months
  The PSP Scale is completed by the physician. PSP is a rating of a patient's level of functioning during the past month in 4 areas: (a) socially useful activities (including work and study); (b) personal and social relationships; (c) self-care; and (d) disturbing and aggressive behaviors. Scores range from 1 to 100. (1= Lack of autonomy in basic functioning and 100 = Excellent functioning in all 4 main areas).
Change from baseline to 24 months in Strauss-Carpenter Levels of Function (LOF) scores | Baseline to 24 months
  The Strauss-Carpenter LOF is completed by the physician. It consists of 9 items that can be grouped into 4 subscales: symptoms (absence of symptoms and recent hospitalizations), social contacts (frequency and quality of social contacts), work (quantity and quality of useful work), and function (ability to meet basic needs, fullness of life, and overall level of function). Each item is rated on a scale of 0 (worst functioning) to 4 (best functioning).

SECONDARY OUTCOMES:
Change from baseline to 24 months in Quality of Life Assessment: Medical Outcomes Survey Short Form (SF-36) scores | Baseline to 24 months
  Patients completed the SF-36. The survey includes 36 items and evaluates health status in the past 4 weeks, in 8 different areas, which can be broadly summarized as physical health (physical functioning [PF], role-physical [RP], bodily pain [BP] and general health [GH]) and mental health (vitality [VT], social functioning [SF], role-emotional [RE], and mental health [MH]). In addition, the SF-36 evaluates health status in 2 broadly-defined areas, mental health and physical health. Higher scores represent better health status.
Change from baseline to 24 months in patient satisfaction with antipsychotic medication | Baseline to 24 months
  Patients are asked a single question to evaluate patient satisfaction with their current Anti psychotic medication. The question is, "The way I feel about my current antipsychotic is:" and used a 7-point response scale from 1 to 7 (extremely dissatisfied to extremely satisfy).
Change from baseline to 24 months in healthcare resource utilization | Baseline to 24 months
  Healthcare resource utilization including dates of hospitalizations (inpatient), emergency room (ER) visits, and outpatient visits, consultations with specialists and general practitioners. Relapse rates (from psychiatric hospitalizations, suicidal behavior or homicidal behavior) are also captured as resource utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP
Locations (1):
- Rockville, Maryland, United States

REFERENCES:
- [Derived] Crivera C, DeSouza C, Kozma CM, Dirani RD, Mao L, Macfadden W. Resource utilization in patients with schizophrenia who initiated risperidone long-acting therapy: results from the Schizophrenia Outcomes Utilization Relapse and Clinical Evaluation (SOURCE). BMC Psychiatry. 2011 Oct 14;11:168. doi: 10.1186/1471-244X-11-168. PMID 21999370
- [Derived] Macfadden W, DeSouza C, Crivera C, Kozma CM, Dirani RD, Mao L, Rodriguez SC. Assessment of effectiveness measures in patients with schizophrenia initiated on risperidone long-acting therapy: the SOURCE study results. BMC Psychiatry. 2011 Oct 14;11:167. doi: 10.1186/1471-244X-11-167. PMID 21999346
- [Derived] Lambert T, Olivares JM, Peuskens J, DeSouza C, Kozma CM, Otten P, Crivera C, Jacobs A, Macfadden W, Mao L, Rodriguez SC, Dirani R, Akhras KS. Effectiveness of injectable risperidone long-acting therapy for schizophrenia: data from the US, Spain, Australia, and Belgium. Ann Gen Psychiatry. 2011 Apr 4;10:10. doi: 10.1186/1744-859X-10-10. PMID 21463526
- See also: The SOURCE Study: Schizophrenia Outcomes-Utilization, Relapse, and Clinical Evaluation — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=348&filename=CR005035_CSR.pdf